CLINICAL TRIAL: NCT06793410
Title: Vaccination Against Human Papillomavirus (HPV) in Women and Men After Stem Cell Transplantation
Brief Title: Vaccination Against Human Papillomavirus (HPV) After Allogeneic Stem Cell Transplantation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ALLO-HPV
Record Dates: First submitted 2025-01-13; First posted 2025-01-27 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Recipients of Allogeneic Stem Cell Transplantation; HPV (Human Papillomavirus)-Associated; Acute Myeloid Leukaemia; Myelodysplastic Syndrome; Diffuse Large B Cell Lymphoma (DLBCL)
MeSH Terms: conditions — Papillomavirus Infections; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Lymphoma, Large B-Cell, Diffuse | interventions — Human Papillomavirus Recombinant Vaccine nonavalent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Late vaccination group (Active Comparator): Subjects will receive Gardasil 9® as part of the late post-transplant vaccination, starting at 15 months after stem cell transplantation.
  Interventions: Biological: Late post-transplant vaccination with Gardasil 9®
- Early vaccination group (Experimental): Subjects will receive Gardasil 9® as part of the early post-transplant vaccination, starting at 9 months after stem cell transplantation.
  Interventions: Biological: Early start post-transplant vaccination with Gardasil 9®

INTERVENTIONS:
Biological: Early start post-transplant vaccination with Gardasil 9® — Subjects will receive Gardasil 9® as part of the early post-transplant vaccination, starting at 9 months after transplantation.
  Arms: Early vaccination group
Biological: Late post-transplant vaccination with Gardasil 9® — Subjects will receive Gardasil 9® as part of the late post-transplant vaccination, starting at 15 months after stem cell transplantation.
  Arms: Late vaccination group

SUMMARY:
Patients who undergo allogeneic stem cell transplantation lose previously acquired immunity and are routinely revaccinated against many infectious diseases. For several reasons, these patients have a long-term immune deficiency due to the transplant itself (lack of immune reconstitution) and due to possible complications, primarily GvHD and its treatment. The risk of secondary malignancy in the long-term following an allogeneic bone marrow transplant is greatly increased, and secondary cancer cases account for a significant proportion of late deaths in both women and men after transplantation. Some of these secondary cancers are associated with HPV. The risk of cervical cancer has been reported to be 13 times increased compared to a healthy population.

Therefore in this trial, the aim is to study immune response (antigen-specific antibody response) after vaccination with 9-valent HPV vaccine (Gardasil 9®) in adult women and men (up to and including 45 years of age) who have undergone allogeneic stem cell transplantation. In this trial, the sponsor will compare "early" (start 9 months after tx) with "late" (start 15 months after tx) vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of AlloSCT from related or unrelated donor.
* Adults (men and women) ≥18 years up to and including 45 years of age for vaccination.
* Patients can be included regardless of prior HPV vaccination prior to transplantation

Exclusion Criteria:

* Severe thrombocytopenia (under 50 x 10^9) not allowing intramuscular injection
* Severe acute GvHD grade III-IV.
* Extensive chronic GvHD requiring treatment with prednisone doses above 0.7 mg/kg/day plus at least two other systemic treatments against GvHD (for example ruxolitinib or photopheresis).
* Prednisone doses above 1mg/kg/day at study start.
* Treatment with rituximab 6 months before start of vaccination. Doses given later (unusual) do not require exclusion.
* Treatment within 3 months before start of vaccination with iv or sc immunoglobulin.
* Pregnancy, pregnancy desire or active pregnancy planning during time vaccine is given and up to three months after last vaccine dose.
* Treatment with blood thinning medication contraindicating intramuscular injection
* Allergy against Gardasil 9

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2029-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Primary outcome - GMT level against HPV 16 | Early group: at month 16 posttransplant. Late group: at month 22 posttransplant.
  Antibody level (GMT - geometric mean titer) against HPV 16 measured 1 months after the third vaccine dose, early vs late.

SECONDARY OUTCOMES:
Secondary outcome 1 - GMT level against all 9 HPV-serotypes | Early group: at month 16 posttransplant. Late group: at month 22 posttransplant.
  Antibody level (GMT - geometric mean titer) against all 9 HPV-serotypes included in vaccine (-6, -11, -16, -18, -31, -33, -45, -52, -58) measured 1 month after the third vaccine dose. Early vs late.
Secondary Outcome 2 - GMT level against all 9 HPV-serotypes | Early group: at month 27 posttransplant. Late group: at month 33 posttransplant.
  Antibody level (GMT - geometric mean titer) against all 9 HPV-serotypes included in vaccine (-6, -11, -16, -18, -31, -33, -45, -52, -58) measured at 12 months after the third vaccine dose. Early vs late.
Secondary Outcome 3 - Proportion seropositive/negative against 9 HPV-serotypes | Early group: at month 16 and month 27 posttransplant. Late group: at month 22 and month 33 posttransplant.
  Proportion seropositive/negative against 9 HPV-serotypes included in vaccine measured 1 and 12 months after third dose. Early vs late.
Secondary Outcome 4 - Seroconversion against 9 HPV-serotypes | Early group: at month 16 posttransplant. Late group: at month 22 posttransplant.
  Seroconversion against 9 HPV-serotypes included in vaccine, pre-vaccination compared to 1 month after third dose, early vs late.
Secondary Outcome 5 - Proportion seropositive against 7/9 HPV-types | Early group: at month 16 and month 27 posttransplant. Late group: at month 22 and month 33 posttransplant.
  Proportion seropositive against 7/9 HPV-types included in the vaccine at 1 and 12 months after completion of vaccination. Early vs late.

CONTACTS AND LOCATIONS:
Locations (5):
- Sweden (5):
  - Skåne's University Hospital, Lund, Region Skåne
  - Karolinska University Hospital, Stockholm, Region Stockholm
  - Uppsala University Hospital, Uppsala, Region Uppsala
  - Linköping University Hospital, Linköping, Region Östergötaland
  - Sahlgrenska University Hospital, Gothenburg, Västra Götalands Region

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) from this clinical trial will not be publicly shared to protect participant privacy and confidentiality. However, researchers may contact the Principal Investigator to request access to de-identified data.